CLINICAL TRIAL: NCT03628092
Title: Laser Therapy for Vulvovaginal Symptoms in Breast Cancer Patients
Acronym: LAAVA2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LAAVA2
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Vulvovaginal Atrophy; Genitourinary Symptoms and Ill-Defined Conditions
Keywords: genitourinary symptoms of menopause; CO2 fractional ablative laser; Early breast cancer; Vulvovaginal atrophy; Vaginal dryness; Dyspareunia; Vaginal itch; Dysuria
MeSH Terms: conditions — Breast Neoplasms; Dyspareunia; Dysuria

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 Fractional Ablative Laser (Active Comparator): 3 treatments approximately 4 weeks apart with vaginal/vulval laser
  Interventions: Device: CO2 Fractional Ablative Laser
- Placebo (Placebo Comparator): 3 treatments approximately 4 weeks apart with "sham" laser
  Interventions: Device: Placebo

INTERVENTIONS:
Device: CO2 Fractional Ablative Laser — Vaginal / vulval laser treatment
  Other Names: Monalisa Touch; Lotus
  Arms: CO2 Fractional Ablative Laser
Device: Placebo — Sham Device
  Arms: Placebo

SUMMARY:
To determine the efficacy of ablative carbon dioxide laser in the treatment of the signs and symptoms of vulvovaginal atrophy (VVA) or genitourinary syndrome of menopause (GSM) in women with breast cancer.

DETAILED DESCRIPTION:
LAAVA 2 is a double blinded randomised placebo/sham-controlled trial assessing whether fractional ablative carbon dioxide is beneficial in improving symptoms in women with a history of early breast cancer. Patients will be randomly assigned in a 1:1 ratio to either active laser treatment or inactive "sham" laser treatment (setting of close to zero)

Participants will receive the 3 treatments approximately 4 weeks apart. Participants will then be followed up at twelve weeks post completion of treatment and twelve months post completion of treatment. At the twelve week follow up visit, after completion of study procedures, patients will be unblinded and those who received "sham" treatment will be allowed to crossover to "active" treatment if they wish.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of early breast cancer >18 years of age
* At baseline patients must have at least one of five symptoms rated at ≥5 on a 10cm VAS scale. Symptoms include vulvo-vaginal itch, dryness, burning, dysuria and dyspareunia.
* Three groups of patients will qualify:
* Treatment induced premature menopause ≤45 years of age (eg secondary to chemotherapy or oophorectomy) for >6 months
* Premenopausal women on GNRH (gonadotrophin releasing hormone) agonist + tamoxifen or an aromatase inhibitor
* Postmenopausal women on tamoxifen or an aromatase inhibitor
* Willingness to give written informed consent and willingness to comply with the study
* Up to date pap test / HPV (human papillomavirus) testing

Exclusion Criteria:

* Medical contraindication to the use of fractional ablative CO2 laser
* Use of oestrogen therapies (systemic or local) in the 6 weeks prior to study treatment
* Use of vaginal lubricants or moisturisers 14 days prior to the study treatment
* Active or recent genitourinary infections (<30 days)
* Genital prolapse (grade III)
* Active or symptomatic vulvo-vaginal dermatological conditions (Lichen sclerosus, lichen planus, vulval psoriasis, Chron's disease, Hidradenitis Suppurativa, vulval dermatitis, candida, chronic vulvovaginal candidiasis, vulval intraepithelial neoplasia, genital warts)
* Inability to tolerate the use of fractional ablative CO2 laser (eg vaginismus)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal dryness | 12 weeks after completion of treatment
  Improvement in vaginal dryness on a 10cm visual analog scale (VAS). A 10cm VAS is a scale from 0 to 10 with 0 being no symptoms and 10 being worst symptoms possible.

SECONDARY OUTCOMES:
Other symptoms of vulvovaginal atrophy | 12 weeks after completion of treatment and 12 months after active treatment
  Improvement in itch, burning, dysuria, dyspareunia and urinary incontinence of a 10cm visual analog scale (VAS)
Maturation index | 12 weeks after completion of treatment and 12 months after active treatment
  Improvement in maturation index from a vaginal swab (a pathological test: the maturation index counts 200 cells and compares the ratio of parabasal:intermediate:superficial squamous cells. Oestrogen deficient smears will show fewer superficial cells and an increase in parabasals (implies an atrophic picture)
  )
Vaginal pH | 12 weeks after completion of treatment and 12 months after active treatment
  Improvement in vaginal pH
Clinician Assessed Changes | 12 weeks after completion of treatment and 12 months after active treatment
  Improvement in vaginal moistness, colour and labia stickiness (moistness and stickiness assessed by a physician as present or not, colour as assessed on a predefined colour chart out of 4 colours).
Quality of Life (QOL) of patients assessed on the Vulval Quality of Life Index | 12 weeks after completion of treatment and 12 months after active treatment
  Improvement in QOL assessed on the Vulval Quality of Life Index (VQLI) -a validated tool. The scoring bands of the VQLI includes: 0-5 = no effect on patient's life, 6-13 = small effect on patient's life, 14-23 = moderate effect on patient's life, 24-37 = very large effect on patient's life, 38-45 = extremely large effect on patient's life.
Sexual Function | 12 weeks after completion of treatment and 12 months after active treatment
  Improvement in sexual function assessed on the Female Sexual Function Index (FSFI) - a validated tool
Satisfaction with treatment assessed on a Likert Scale | 12 weeks after completion of treatment and 12 months after active treatment
  Patient satisfaction assessed on Likert Scale - a validated tool scoring from 1 to 5 (1=strongly disagree, 2=disagree, 3= neutral, 4=agree, 5=strongly agree)
Safety of laser treatment (Side effects) | 15 months
  Side effects reported over the duration of the study will be collected descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Pearson, BMed, Principal Investigator — Royal North Shore Hospital
Locations (2):
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales